CLINICAL TRIAL: NCT02709603
Title: Randomized Clinical Trial of Oral Hyoscine Butyl Bromide in Reducing Pain During HSG
Brief Title: Hyoscine Butyl Bromide in Reducing Pain During HSG
Acronym: HBTB-DIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HS2
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Pain Relief With HSG
MeSH Terms: interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): oral hyoscine butyl bromide; 2 tablets (buscopan 10 mg) 30 minutes before the procedure
  Interventions: Drug: hyoscine butyl bromide
- Group B (Placebo Comparator): oral 2 tablets (PLACEBO) 30 minutes before the procedure
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: hyoscine butyl bromide — oral hyoscine butyl bromide; 2 tablets (buscopan 10 mg) 30 minutes before the procedure
  Other Names: BUSCOPAN
  Arms: Group A
Drug: placebo — oral placebo; 2 tablets 30 minutes before the procedure
  Arms: Group B

SUMMARY:
Many oral analgesic drugs such as nonsteroidal anti-inflammatory drug(NSAID) are used to relieve pain from gynecological procedure and dysmenorrhea. Hyoscine-N-butyl bromide, an antispasmodic drug are commonly used for relief of smooth muscle spasms and can use to relieve genito-urinary spasm. Some studies reported hyoscine can't relieve pain in minor gynecological procedures. So the efficacy of hyoscine use are still controversial and no previous studies investigated its efficacy for pain relief in HSG procedure.

ELIGIBILITY:
Inclusion Criteria:

The infertile women who indicated for HSG.

Exclusion Criteria:

* contraindications to Hyoscine or NSAID - known sensitivity to these drugs
* known sensitivity to contrast media
* abnormal uterine bleeding
* genital tract infection
* suspected pregnancy

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean pain score during. hysterosalpingography by visual analog scale | intraoperative

SECONDARY OUTCOMES:
Mean pain score after hysterosalpingography | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abbas, MD, Principal Investigator — Woman health hospital Assiut
Locations (2):
- Egypt (2):
  - Ahmed Abbas, Assiut, Cairo Governorate
  - Ahmed Abbas, Asyut, Please Select

IPD SHARING:
Plan to Share IPD: Undecided